CLINICAL TRIAL: NCT03368365
Title: Validation of the Rest Respiratory Function Monitoring of Pulmonary Transplants at Home to Anticipate Unplanned Hospitalizations
Brief Title: Validation of the Respiratory Function of Pulmonary Transplants to Anticipate Unplanned Hospitalizations
Acronym: TRANSADOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Aqsitania SAS (Unknown); AGIR à Dom (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 38RC16.132; 2016-A01060-51 (Registry Identifier: Agence National de Sécurtié du Médicament (ANSM)); 16-CHUG-17 (Registry Identifier: Comité de Protection des Personnes (CPP) Sud-Est V)
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Lung Transplant; Complications
Keywords: Monitoring; Home; Lung; Transplant; Hospitalization; Respiratory function at rest; Monitoring modem

STUDY DESIGN:
Intervention Model Description: All transplanted subjects will be equiped with the Ventilotel (r) after their inclusion in the study.
Masking Description: The occurrence of unplanned hospitalizations is independent of the spirometer used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ventilotel ® (Other): Using of the spirometer of Aqsitania company, Ventilotel ®.
  Interventions: Device: Ventilotel ®

INTERVENTIONS:
Device: Ventilotel ® — Using of the spirometer of Aqsitania company, Ventilotel ®, to analyse the respiratory function at rest and to predict unplanned hospitalizations.

SUMMARY:
Acute cellular and/or humoral rejection and early graft infections after pulmonary transplant (<2.5 years) are common and can lead to chronic dysfunction of the transplanted organ or Chronic Lung Allograft Dysfunction, CLAD. These complications increase the number of unplanned and life-threatening hospitalizations. Regular multi-weekly monitoring of respiratory function is necessary to detect these complications early and to make their management more effective and less costly. Monitoring by micro spirometers with forced expirations at home proved difficult to perform (patient and effort dependent), often poorly coordinated (transmission of data to practitioners) and not sensitive in the prediction of post-transplant complications. Aqsitania has developed an innovative analysis of resting respiratory signals. This innovative analysis is called "Anharmonic Morphological Analysis of Respiratory Signals (AMARS)". This automated analysis is based on a measurement of the respiration collected by a spirometry device communicating and allowing a remote home monitoring (Ventilotel®). We hypothesize that this Anharmonic Morphological Analysis of Respiratory Signals at rest could predict unplanned hospitalizations and allow for more reliable monitoring of pulmonary transplant patients. Inclusion visit: Explanation of the study and collection of consent, measurement of resting breath and explanation on the mode of use of the measuring device at home, clinical examination, respiratory functional exploration. Follow-up at home for 12 months with a resting breath measurement for 2 to 3 min, in the morning on waking and in the evening before bed, 2 days / week with automatic sending of data on the Aqsitania server. The first month, a visit at home can be made if the subject feels the need. At each measurement, Aqsitania transmits the data in the e-CRF, a report that gives the anonymised values of the markers and the current personal respiratory profile. In order to avoid "motivational" bias, patients will have instructions to use the device but no "coaching" call will be made during the study. Patients will have their monthly or quarterly follow-up visits, including clinical examination, respiratory functional exploration and an analysis of adverse events. No additional search-specific visits will be carried out.

DETAILED DESCRIPTION:
Acute cellular and/or humoral rejection and early graft infections after pulmonary transplant (<2.5 years) are common and can lead to chronic dysfunction of the transplanted organ or Chronic Lung Allograft Dysfunction, CLAD. These complications increase the number of unplanned and life-threatening hospitalizations. Regular multi-weekly monitoring of respiratory function is necessary to detect these complications early and to make their management more effective and less costly. Monitoring by micro spirometers with forced expirations at home proved difficult to perform (patient and effort dependent), often poorly coordinated (transmission of data to practitioners) and not sensitive in the prediction of post-transplant complications. Aqsitania has developed an innovative analysis of respiratory signals at rest. This innovative analysis is called "Anharmonic Morphological Analysis of Respiratory Signals (AMARS)". This automated analysis is based on a measurement of the respiration collected by a spirometry device communicating and allowing a remote home monitoring (Ventilotel®). We hypothesize that this Anharmonic Morphological Analysis of Respiratory Signals at rest could predict unplanned hospitalizations and allow for more reliable monitoring of pulmonary transplant patients.

Individual benefit (s): From an individual point of view, this is a descriptive study with no direct benefit expected for the patients participating in the research. Nevertheless, if the hypothesis is confirmed, the benefits for the transplant patients will be considerable because a prediction of the occurrence of post-transplant complications at a much earlier stage, probably infra-clinical, would allow a more efficient management thus a better prognosis for these patients grafted. This is added the advantage of the telecommunication system which will allow a reliable and automated transmission of the parameters evaluated at home, which can improve the coordination of the care and the reactivation of the caregivers. Lastly, it is possible to emphasize the medical and psychological safety of the patient by the use of this device, which is an important element for this type of risky situation.

Collective Benefit (s): Provided that subsequent randomized studies confirm this, it is likely that monitoring of respiratory function by this innovative connected device will significantly reduce the morbidity and mortality of post-transplant follow-up. Collective benefits are also economic. Significant savings in the use of care and hospitalizations avoided or reduced in anticipation of the risk of serious complications following pulmonary transplantation can be expected from this new mode of surveillance. The challenge would be to significantly increase the cost effectiveness of this costly therapeutic in 2015 to eventually have a QALY <100 000 €.

Expected benefits: If the analysis of respiration at home allows prediction of complications after a pulmonary transplant, it will then be necessary to demonstrate that an early management strategy, probably subclinical and based on this analysis, Avoid post-transplant complications, reduce morbidity and mortality and care for pulmonary transplant patients. The results for this research are therefore considerable.

Medical device used in research:

The device used for home monitoring of respiratory function of pulmonary transplant patients will be Ventilotel®, developed by Aqsitania and manufactured by Thor Medical Systems, an internationally recognized manufacturer of this type of equipment. This device is marked CE and class IIa. Ventilotel® is a communicating device for measuring the respiratory function of a patient in calm ventilation. The measure consists in breathing a patient by the mouth, for about 3 minutes in a ventilometer, the nose blocked by a nose clip. The measure taken is transmitted, anonymised, by the GSM 3G network to Aqsitania's digital analysis platform for the signal processing and the calculation of the associated markers. Then the platform sends the data directly into the e-CRF. The Ventilotel® is composed of 3 main parts: 1. a USB ultrasonic ventilometer or pneumotachograph, intended for the measurement itself (2 hull variants: reinforced with silicone, or light). The white plastic tube through it is the place where the patient will breathe, protected by an antiviral / antibacterial filter to change every month. 2. a computer case for controlling the ventilometer and for transmitting the acquired information to the remote signal analysis platform. 3. a USB barcode reader, designed to read the barcode of the patient's paper file, to perform a measurement for which it is desired to request a calculation of the Aqsitania bio-markers. It comes with a USB port reducer for use with the computer case.

Patient Selection:

In the month preceding a scheduled hospitalization for assessment, the investigating physician validates the first eligibility criteria based on the patient's medical record. In case of eligibility, the CRA calls the patient to inform him / her of the possible participation in the protocol and gives an initial information on the protocol. He sends him the information note by post with a delay of at least a week between the receipt of the mail and the planned hospitalization. During the hospitalization scheduled for assessment, the investigating physician re-informs the patient and answers all his questions concerning the objective, the nature of the constraints, the foreseeable risks and the expected benefits of the research. It also specifies the rights of the subject in the context of biomedical research. The investigating physician is responsible for obtaining the informed informed consent of the subject. The consent form must be signed prior to any clinical or paraclinical examination required by the research.

Inclusion Visit:

Obtaining consent: If the participant gives his / her participation agreement, the participant and the investigator enter their first and last names in clear, date and sign the consent form in two original copies. The different copies of the information memorandum and the consent form are then distributed as follows: a copy of the information memorandum and the signed consent is given to the subject, the other copy is retained by the investigating physician in a place Inaccessible to third parties. At the end of the inclusions or at the latest at the end of the search, a copy of each consent form shall be forwarded to the proponent or its representative according to procedures communicated to investigators in a timely manner.

Conduct of the visit: The inclusion visit, provided by the investigating physician, includes:

* Clinical examination: weight, height, temperature, blood pressure, pulse rate, respiratory rate, pulmonary auscultation.
* Spirometry with Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC), Forced Expiratory Flow between 25 and 75% of FVC (FEF 25-75), Functional Residual Capacity (FRC), the Total Lung Capacity (TLC), the Residual Volume (VR) and the Expiratory Reserve Volume (ERV).
* A measure of peak expiratory flow (PEF).
* A demonstration of the use of the instrument for measuring spontaneous breathing parameters (Ventilotel®, Aqsitania) as well as its putting into operation: at the inclusion visit, the casing is connected momentarily to the barcode reader, The patient code is read and stored in the case which will emit measurements with this code,
* A measurement of breathing at rest with Ventilotel® and delivery of the device to the patient.

Follow-up visits:

Follow-up visits will be done at the usual rythm defined for each patient according to the age of his or her transplant or his / her status (usually: monthly visits the first post-transplant year, quarterly the second year). These visits will be in accordance with the usual follow-up except for an additional measure carried out with the Ventilotel®.

Measures at home:

At the patient's home, the patient will be asked to measure breathing at rest with Ventilotel® in the morning and evening, twice a week and for 1 year. During the first month, a visit to the patient's home can be made if the patient feels the need to assist in the handling of Ventilotel®. The measure consists of breathing through the mouth, for about 3 minutes in the ventilometer, the nose blocked by a nose clip. Then the data is transmitted to the Aqsitania servers, which will send the data directly to the e-CRF. If the GSM signal is temporarily lost during the measurement, the Ventilotel® can store the respiratory data and send it to Aqsitania later when the GSM signal is returned. During a week without data transmission, the CRA referent of the site from which the patient is born will call Aqsitania in order to know if the box is connected to the network. In this case, the absence of data will result from a non-observance of the patient at Ventilotel® and nothing will be done in addition. If, on the contrary, the Ventilotel® appears to be disconnected from the Aqsitania servers, a call will be sent to the patient in order to know if he has disconnected the device because it no longer uses it or if it has broken down . If it is unplugged, nothing will be done. If it fails (device plugged in but does not start or does not transmit data despite good network quality), a home visit will be made by the CRA to simply replace the defective hardware (without motivate the patient to use the device). The patient continues to use the Spirotel provided after the transplant as recommended by the transplant team. The Spirotel is a mini-spirometer for measuring Forced Vital Capacity (FVC), Forced Expiratory Volume in 1 second (FEV1) and FEV1/FVC (forced maneuvers).

End search visit:

The end-of-study visit at 12 months will correspond to the closest visit of 12 months programmed in the usual follow-up of the patient. It will include:

* Clinical examination: weight, height, temperature, blood pressure, pulse rate, respiratory rate, pulmonary auscultation.
* Spirometry with Forced Expiratory Volume in 1 second (FEV1), Forced Vital Capacity (FVC), Forced Expiratory Flow between 25 and 75% of FVC (FEF 25-75), Functional Residual Capacity (FRC), the Total Lung Capacity (TLC), the Residual Volume (VR) and the Expiratory Reserve Volume (ERV).
* A measure of Peak Expiratory Flow (PEF).
* A measure of resting breathing with Ventilotel® and delivery of the device to the CRA referent of the study on the site.

Compendium of unplanned hospitalizations:

Any hospitalization additional to the schedule of hospitalizations scheduled for follow-up will be considered as an unplanned hospitalization. All causes of unplanned hospitalization will be retained. The causes of unscheduled hospitalizations will be reported in the hospitalization reports. Consultations (programmed or not) will not be included in the primary endpoint.

AMARS Settings:

The 8 "morphological" Aqsitania markers characterizing breathing at rest are:

4 parameters measured at "inspiratory" times

* A1 Amplitude of the inspiratory front
* B1 Asymmetry of the inspiratory front
* R1 Anharmonicity of the inspiratory front
* T1 Position of the inspiratory front 4 parameters measured at expiratory times
* A2 Amplitude of the expiratory front
* B2 Asymmetry of the expiratory front
* R2 Anharmonicity of the expiratory front
* T2 Position of the expiratory front

These 8 parameters are evaluated on each of the breathing cycles at rest of a set of 30 to 50 consecutive respiratory cycles measured from 2 to 3 minutes on a day in the morning and evening. The mean value and the standard deviation of each morphological parameter are evaluated on this set of cycles. The reference values of these 8 parameters are determined for each patient during the inclusion visit. The results of each measure at home are expressed in absolute values and in percentage of variation compared to the reference values. These 8 parameters are analyzed alone or combined at different times before each event. In addition to the 8 specific parameters, the tidal volume and respiratory rate are also measured as well as the stability of the Personal Respiratory Profile. The AMARS parameters and the unplanned hospitalizations will be coded independently in the e-CRF: the AMARS parameters will be automatically transferred to the e-CRF; Hospitalizations coded by a clinical research associate. The statistical analysis will be carried out after the database has been frozen and the statistician who analyzes the data will not have participated in the coding of the events.

Statistical aspects:

1. Graphical analysis of the evolution of the parameters of breath at rest according to the occurrence of unplanned hospitalizations:

   * per patient,
   * overall.

   This graphical analysis will be performed for each of the 8 parameters of normal breathing as well as for some parameter associations. This step will identify which parameters or associations of parameters fluctuate according to the occurrence of unplanned hospitalizations (predictive power), as well as the time in days between the fluctuation of the parameter and the hospitalization.
2. ROC curve analysis: These ROC curves will be performed only for parameters or parameters associations that have shown a predictive power in step 1. The ROC curves will determine the threshold of discrimination of the parameters or combination of parameters which provides the best sensitivity and the best specificity for the prediction of hospitalizations. The PPV and NPV will also be determined. Internal validation using a bootstrap technique will be carried out. This internal validation will make it possible to evaluate the optimism bias. A calibration will be performed by a Hosmer-Lemeshow analysis or another suitable model.
3. Analysis of ANOVA variance and Bonferroni test: This step will be performed only for parameters or associations of parameters that have shown a predictive power in step 1. ANOVA will identify factors influencing parameters or associations of parameters such as the severity of bronchiolitis obliterans syndrome or restrictive impairment.
4. Calculation of the correlation coefficients (Pearson or Spearman coefficient, depending on whether the variables follow a normal distribution) between the parameters of classical spirometry and those of respiration at rest.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female, pulmonary transplant for at least three months but less than 2.5 years in stable condition (absence of unplanned hospitalization, antibiotic treatment or modification of treatment during the month preceding inclusion).
* Having given informed consent in writing and affiliated to a social security scheme.

Exclusion Criteria:

* Home network coverage insufficient for data transmission.
* Proven psychiatric pathology.
* Cognitive problem significantly limiting the understanding of different instructions or evaluations.
* People referred to Articles L1121-5 to L1121-8 of the Code of Public Health.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Analyze AMARS parameters to predict unplanned hospitalizations. | 12 months
  Criterion including Sensitivity (Se), Specificity (Sp), Positive Predictive Value (VPP) and Negative Predictive Value (VPN) of AMARS parameters to predict unplanned hospitalization with measurement of the delay between changes in respiration at rest and unplanned hospitalization.

SECONDARY OUTCOMES:
Compare spirometry carried out at home and that performed in consultation / hospitalizations. | 12 months
  Correlation between standard FEV1, FVC (estimated by spirometry and micro-spirometry) and AMARS parameters.
Determine the diagnostic specificities of the AMARS Analysis | 12 months
  Analysis of factors influencing AMARS parameters such as types of complications: acute rejection, opportunistic infections, proximal bronchial complications.
Analyze the feasibility of pulmonary function monitoring at home by the Ventilotel (r) device in pulmonary transplant patients. | 12 months
  Percentage of patients able to perform resting breath measurement for 2 to 3 minutes on waking and before bed, at least twice a week and for 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Pison, Pr MD PhD, Principal Investigator — University Hospital, Grenoble; Jean-Christian Borel, PhD, Study Chair — AGIR à Dom; José Labarère, Pr PhD, Study Chair — Clinical Investigation Center - Technological Innovation (CIC-Innovation Technologique)
Locations (2):
- France (2):
  - Grenoble University Hospital, La Tronche, Auvergne-Rhône-Alpes
  - Lyon University Hospital, Lyon, Rhônes-Alpes

IPD SHARING:
Plan to Share IPD: No